CLINICAL TRIAL: NCT01412294
Title: Phase II Study to Evaluate Efficacy and Safety of Capecitabine/Cisplatin Combination Therapy in Gastric Cancer Patients Who Relapsed After S-1 Adjuvant Chemotherapy (XParTS)
Brief Title: XParTS: Capecitabine/Cisplatin(XP) for Recurrent Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRIN-GC1106-XParTS; UMIN000005857 (Other: UMIN Clinical Trials Registry)
Record Dates: First submitted 2011-07-30; First posted 2011-08-09 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; recurrent gastric cancer; adenocarcinoma of the stomach; capecitabine; xp
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, Cisplatin (Experimental)
  Interventions: Drug: Capecitabine, Cisplatin

INTERVENTIONS:
Drug: Capecitabine, Cisplatin — Drug: Capecitabine Capecitabine will be administered at 1,000 mg/m2 orally, twice daily (2,000 mg/m2 total daily dose) on Days 1 through 14 of each 21-day treatment cycle.
  Drug: Cisplatin Cisplatin will be administered at 80 mg/m2 by intravenous infusion on Day 1 of each 21-day treatment cycle.

SUMMARY:
The aim of this study is to evaluate efficacy and safety of Capecitabine/Cisplatin for gastric cancer patients who relapsed after adjuvant chemotherapy by S-1.

DETAILED DESCRIPTION:
S-1/Cisplatin (SP) is one of the standard treatments of advanced gastric cancer. However, evidence of SP on gastric cancer recurrence after adjuvant therapy by the same drug (S-1) is not established. The aim of this study is to evaluate the efficacy and safety of Capecitabine/Cisplatin (XP) for gastric cancer patients who relapsed after adjuvant chemotherapy by S-1.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent gastric cancer histologically confirmed as being adenocarcinoma
2. Age of 20 to 74 years with either gender
3. ECOG Performance Status of 0 to 2
4. Lesions confirmed on imaging within 28 days before registration (not required measurable lesions as defined in RECIST version 1.1)
5. Post-gastrectomy adjuvant chemotherapy including S-1 for at least 12 weeks including interruption period
6. Less than 6 months treatment-free interval from completion of adjuvant therapy
7. In case with receiving neoadjuvant chemotherapy, the total dose of CDDP does not exceed 120mg/m2
8. Treatment-naïve recurrent gastric cancer
9. Life expectancy of at least 3 months after registration
10. Written informed consent
11. Adequate major organ functions within 14 days before registration

    Exclusion Criteria:
12. Positive HER2 status
13. Previous treatment with platinum agents after curative surgery
14. Previous history of serious hypersensitivity to fluoropyrimidines or platinum agents
15. Previous history of adverse reactions suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency
16. More than one cancer at the same time or more than one cancer at different times separated by a 5-year disease-free interval. However, multiple active cancers do not include carcinoma in situ or skin cancer which is determined to have been cured as a result of treatment.
17. Obvious infection or inflammation (pyrexia ≥ 38.0˚C)
18. Active hepatitis
19. Heart disease that is serious or requires hospitalization, or history of such disease within past year

9) Concurrent illness that is serious or requires hospitalization (intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, poorly controlled diabetes mellitus, renal failure, liver disorders, or hepatic cirrhosis)

10) Being treated or in need of treatment with phenytoin or warfarin potassium

11) Chronic diarrhea (watery stool or ≥ 4 times/day)

12) Active gastrointestinal hemorrhage

13) Body cavity fluids requiring drainage or other treatment

14) Clinical suspicion or previous history of metastases to brain or meninges

15) Women who are pregnant, breastfeeding, or potentially (hoping to become) pregnant 16) Unwillingness to practice contraception

17) Poor oral intake

18) Psychiatric disorders which are being or may need to be treated with psychotropics

19) Otherwise determined by investigators or site principal investigators to be unsuitable for participation in study

Ages: 20 Weeks to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 year

SECONDARY OUTCOMES:
Overall survival | 2 year
Response rate | 2 year
Time to treatment failure | 2 year
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Akira Tsuburaya, Principal Investigator — Shonan Kamakura Hospital
Locations (1):
- Epidemiological and Clinical Research Information Network, Kyoto, Japan

REFERENCES:
- [Derived] Nishikawa K, Tsuburaya A, Yoshikawa T, Takahashi M, Tanabe K, Yamaguchi K, Yoshino S, Namikawa T, Aoyama T, Rino Y, Kawada J, Tsuji A, Taira K, Kimura Y, Kodera Y, Hirashima Y, Yabusaki H, Hirabayashi N, Fujitani K, Miyashita Y, Morita S, Sakamoto J. A phase II trial of capecitabine plus cisplatin (XP) for patients with advanced gastric cancer with early relapse after S-1 adjuvant therapy: XParTS-I trial. Gastric Cancer. 2018 Sep;21(5):811-818. doi: 10.1007/s10120-018-0815-0. Epub 2018 Feb 27. PMID 29488122